CLINICAL TRIAL: NCT06340464
Title: Investigation & Comparison of the Effects of Preoperative Nutritional Status Scores to Predict Post-op Pulmonary Complications Among Elderly Patients With Cardiac Surgery
Brief Title: Preoperative Nutritional Status Scores to Predict PPC in Elderly With Cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Panalee Kittisopaporn, Miss, Prince of Songkla University
Other Study IDs: REC.67-018-8-1
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Cardiac Surgery; Elderly Patient; Postoperative Pulmonary Complication; Nutrition Scoring System
Keywords: Cardiac surgery; Elderly, Aged; Postoperative pulmonary complication; Nutrition scoring system; GNRI; MNA; PNI
MeSH Terms: interventions — Serpin E2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: GNRI, PNI, MNA — Nutrition scoring systems

SUMMARY:
This prospective study investigate prognostic values and compare the role of nutritional status by using GNRI, MNA, and PNI in predicting post-operative pulmonary complication among elderly patients with cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patient age ≥ 60 years
* Open heart surgical procedure on pump (CABG, valvular disease, combine CABG and valve surgery
* Elective surgery

Exclusion Criteria:

- Emergency surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly patients (aged ≥ 60 years old) who undergoing cardiac surgery in Songklanagarind hospital, Songkla, Thailand
Sampling Method: Non-Probability Sample
Enrollment: 229 (Estimated)
Dates: Start 2024-03-21 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pulmonary complication | 1 month
  PPCs such as pneumonia, pulmonary embolism, ventilation longer than 24 h, pleural effusions necessitating drainage and reintubation within 72 h of extubation

CONTACTS AND LOCATIONS:
Overall Officials: Panalee Kittisopaporn, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Prince of Songkla University
Locations (1):
- Department of Anesthesiology, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand